CLINICAL TRIAL: NCT06703710
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose, Phase 1 Clinical Trial to Evaluate the Safety/Tolerability and PK Characteristics, and to Explore Food Effect and Ethnic Difference of JW2286 in Healthy Volunteers
Brief Title: To Evaluate the Safety/Tolerability and Pharmacokinetic Characteristics in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: JW23104
Record Dates: First submitted 2024-11-18; First posted 2024-11-25 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group (JW2286) (Experimental): Ethnicity: Korean or Caucasian
  Interventions: Drug: JW2286
- Placebo group (Placebo of JW2286) (Placebo Comparator): Ethnicity: Korean or Caucasian
  Interventions: Drug: Placebo of JW2286

INTERVENTIONS:
Drug: JW2286 — a single administration of JW2286 per dose
  Arms: Test group (JW2286)
Drug: Placebo of JW2286 — a single administration of Placebo of JW2286 per dose
  Arms: Placebo group (Placebo of JW2286)

SUMMARY:
This clinical trial is a randomized, double-blind, placebo-controlled, single ascending dose, phase 1 clinical trial to evaluate the safety/tolerability and pharmacokinetic characteristics, and to explore food effect and ethnic difference of JW2286 after oral administration in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Korean or Caucasian volunteers

Exclusion Criteria:

* Individuals with a clinically significant disease or history
* Individuals with a history of a gastrointestinal disorder or surgery
* In the case of all female individuals with childbearing potential, except for those who are surgically sterile

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve from 0 to last (AUClast) of JW2286 | 0 to 168 hours
  Pharmacokinetic Characteristics Evaluation
Area under the plasma drug concentration-time curve from 0 to infinity (AUCinf) of JW2286 | 0 to 168 hours
  Pharmacokinetic Characteristics Evaluation
The maximum or peak concentration between zero and dosing interval (Cmax) of JW2286 | 0 to 168 hours
  Pharmacokinetic Characteristics Evaluation
Time of Maximum Concentration (Tmax) of JW2286 | 0 to 168 hours
  Pharmacokinetic Characteristics Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No